CLINICAL TRIAL: NCT07217691
Title: Optimization of Commissural Alignment During Transcatheter Aortic Valve Implantation With Evolut FX+. A Randomized, Prospective Study.
Brief Title: Optimization of Commissural Alignment During Transcatheter Aortic Valve Implantation With Evolut FX+
Acronym: ALIGN-EFX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Al-Ani, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 904586
Record Dates: First submitted 2025-09-23; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Aortic Stenosis; Trans-catheter Aortic Valve Implantation; Commissural Alignment
Keywords: TAVI; Commissural alignment
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard rotation of delevery system in the descending aorta at LAO 25 degree (Active Comparator): LAO 25
  Interventions: Device: Implantation of Evolut FX pluss TAVI device from Medtronic in LAO 25
- Rotation of delivery system in the descending aorta with patient-specific degree obtained from CT (Active Comparator): Patient specific degree
  Interventions: Device: Implantation of Evolut FX pluss TAVI device from Medtronic in patient specific degree.

INTERVENTIONS:
Device: Implantation of Evolut FX pluss TAVI device from Medtronic in LAO 25 — In this arm the HAT marker will be placed in the outer curvature of descending aorta in LAO 25 degree.
  Arms: Standard rotation of delevery system in the descending aorta at LAO 25 degree
Device: Implantation of Evolut FX pluss TAVI device from Medtronic in patient specific degree. — In this arm the HAT marker will be placed in the outer curvature of descending aorta in patient specific degree.
  Arms: Rotation of delivery system in the descending aorta with patient-specific degree obtained from CT

SUMMARY:
Purpose of the Study The purpose of this study is to investigate how a transcatheter aortic valve (TAVI, biological valve prosthesis) can best be positioned in order to avoid blockage of the coronary arteries by the valve material after implantation.

Method The study will include patients undergoing TAVI. Participants will be randomized, meaning that it will be determined by chance which of two established implantation techniques is used. Both techniques are already part of routine clinical practice.

Examinations After the procedure, a CT scan will be performed to evaluate the position of the valve in relation to the coronary arteries. This CT scan is the only additional examination beyond today's standard clinical practice.

Significance If one of the techniques proves to provide better positioning of the valve, this method may be recommended as standard practice in future treatment. The study will therefore contribute to improved patient safety and treatment quality, as well as increase knowledge about optimal positioning and implantation techniques in TAVI.

DETAILED DESCRIPTION:
The purpose of the present study is to prospectively evaluate the efficacy and safety of a novel patient-specific rotation of the Evolut FX+ TAVI valve and the delivering system during the transfemoral (TF) procedure. Specifically, it aims to evaluate and compare the commonly used fluoroscopic (X-ray) LAO degree for rotation of the delivery system and more patient-specific LAO degree achieved by CT analysis prior to the procedure. The degree of alignment and coronary overlap will be measured with ECG-gated CT after the procedure. Thus, it will prospectively explore if these two techniques differ in obtaining commissural alignment, coronary overlap and safety outcomes following implantation of latest-generation Evolut FX+ valve.

We intend to include 40 patients with severe aortic stenosis and in whom TF-TAVI with Evolut FX+ is planned after heart team meeting. Preprocedure CT scan and postprocedure CT scan will be evaluated for commissural alignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe aortic stenosis indicated for TAVI after heart team meeting.
* Age ≥65 years.
* Patients planned by the TAVI team to receive a self-expandable valve (Evolut FX+ valve).
* Patients providing informed consent.

Exclusion Criteria:

* Severe peripheral vascular disease preventing transfemoral access.
* Prior aortic valve replacement or bicuspid valve.
* Severely reduced kidney function (estimated glomerular filtration rate <30).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Achievement commissural alignment. | Day 1 (post-procedure CT).
  Proportion of patients achieving commissural alignment post-TAVI (measured by CT-analysis after TAVI).
Commissural alignment after TAVI measured in degrees. | Day 1 (post-procedure CT)
  Commissural alignment following TAVI, assessed by computed tomography (CT) analysis.
  Native commissures (measured before TAVI from CT) will serve as the reference. We will measure the number of degrees of all three commissures from the center of the left main artery before and after TAVI to estimate alignment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bieliauskas G, Wong I, Bajoras V, Wang X, Kofoed KF, De Backer O, Sondergaard L. Patient-Specific Implantation Technique to Obtain Neo-Commissural Alignment With Self-Expanding Transcatheter Aortic Valves. JACC Cardiovasc Interv. 2021 Oct 11;14(19):2097-2108. doi: 10.1016/j.jcin.2021.06.033. Epub 2021 Sep 15. PMID 34538602
- [Background] Redondo A, Valencia-Serrano F, Santos-Martinez S, Delgado-Arana JR, Barrero A, Serrador A, Gutierrez H, Sanchez-Lite I, Sevilla T, Revilla A, Baladron C, Kim WK, Carrasco-Moraleja M, San Roman JA, Amat-Santos IJ. Accurate commissural alignment during ACURATE neo TAVI procedure. Proof of concept. Rev Esp Cardiol (Engl Ed). 2022 Mar;75(3):203-212. doi: 10.1016/j.rec.2021.02.004. Epub 2021 Mar 26. English, Spanish. PMID 33781722
- [Background] Konami Y, Sakamoto T, Suzuyama H, Horio E, Yamaguchi J. Commissural alignment in the Evolut TAVR procedure: conventional versus hat marker-guided shaft rotation methods. AsiaIntervention. 2023 Sep 21;9(2):156-165. doi: 10.4244/AIJ-D-23-00017. eCollection 2023 Sep. PMID 37736211
- [Background] Tang GHL, Sengupta A, Alexis SL, Zaid S, Leipsic JA, Blanke P, Grubb KJ, Gada H, Yakubov SJ, Rogers T, Lerakis S, Khera S, Adams DH, Sharma SK, Kini A, Reardon MJ. Conventional versus modified delivery system technique in commissural alignment from the Evolut low-risk CT substudy. Catheter Cardiovasc Interv. 2022 Feb;99(3):924-931. doi: 10.1002/ccd.29973. Epub 2021 Oct 9. PMID 34626449
- [Background] Jilaihawi H. When the (Commissural) Stars (Mis)ALIGN. JACC Cardiovasc Interv. 2020 May 11;13(9):1043-1045. doi: 10.1016/j.jcin.2020.03.001. Epub 2020 Mar 16. No abstract available. PMID 32381183
- [Background] Sondergaard L, De Backer O. Transcatheter aortic valve implantation: don't forget the coronary arteries! EuroIntervention. 2018 Jun 20;14(2):147-149. doi: 10.4244/EIJV14I2A24. No abstract available. PMID 29937429
- [Background] Khera S, Krishnamoorthy P, Sharma SK, Kini AS, Dangas GD, Goel S, Lerakis S, Anastasius M, Moreno P, Tang GHL. Improved Commissural Alignment in TAVR With the Newest Evolut FX Self-Expanding Supra-Annular Valve: First-in-Human Experience. JACC Cardiovasc Interv. 2023 Feb 27;16(4):498-500. doi: 10.1016/j.jcin.2022.10.041. Epub 2022 Nov 16. No abstract available. PMID 36858671
- [Background] Tang GHL, Amat-Santos IJ, De Backer O, Avvedimento M, Redondo A, Barbanti M, Costa G, Tchetche D, Eltchaninoff H, Kim WK, Zaid S, Tarantini G, Sondergaard L. Rationale, Definitions, Techniques, and Outcomes of Commissural Alignment in TAVR: From the ALIGN-TAVR Consortium. JACC Cardiovasc Interv. 2022 Aug 8;15(15):1497-1518. doi: 10.1016/j.jcin.2022.06.001. PMID 35926918
- [Background] Fuchs A, Kofoed KF, Yoon SH, Schaffner Y, Bieliauskas G, Thyregod HG, Makkar R, Sondergaard L, De Backer O, Bapat V. Commissural Alignment of Bioprosthetic Aortic Valve and Native Aortic Valve Following Surgical and Transcatheter Aortic Valve Replacement and its Impact on Valvular Function and Coronary Filling. JACC Cardiovasc Interv. 2018 Sep 10;11(17):1733-1743. doi: 10.1016/j.jcin.2018.05.043. Epub 2018 Aug 15. PMID 30121280
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165

DOCUMENTS (1):
  • Study Protocol (2025-10-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT07217691/Prot_000.pdf